CLINICAL TRIAL: NCT04973176
Title: Standard Versus Flexible Tip Bougie for Videolaryngoscopy: A Randomised Comparison Between Standard and Flexible Tip Bougie (Tracheal Tube Introducers) for Tracheal Intubation Using Non Channelled Videolaryngoscope
Brief Title: Standard Versus Flexible Tip Bougie for Videolaryngoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CM538321
Record Dates: First submitted 2021-07-09; First posted 2021-07-22 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endotracheal intubation with C-MAC D Blade Videolaryngoscopy and Standard Bougie (Active Comparator): Patients randomised to standard bougie will be intubated using standard bougie (Frova® airway intubation catheter )
  Interventions: Device: Standard Bougie
- Endotracheal intubation with C-MAC D Blade Videolaryngoscopy and Flexi-tip Bougie (Active Comparator): Patients randomised to Flexi-tio bougie will be intubated using Flexi-tip bougie (P3 medical Ltd, Bristol, UK)
  Interventions: Device: Flexi-tip Bougie (P3 Medical Bristol,UK)

INTERVENTIONS:
Device: Standard Bougie — Standard Bougie for endotracheal intubation
  Arms: Endotracheal intubation with C-MAC D Blade Videolaryngoscopy and Standard Bougie
Device: Flexi-tip Bougie (P3 Medical Bristol,UK) — Flexi-tip Bougie for endotracheal intubation
  Arms: Endotracheal intubation with C-MAC D Blade Videolaryngoscopy and Flexi-tip Bougie

SUMMARY:
This study aims to compare the flexible tip bougie with standard bougie for tracheal intubation using non channelled, acute angled video laryngoscope using modified intubation difficulty scale score as primary outcome.

DETAILED DESCRIPTION:
Videolaryngoscopes are devices which aid successful intubation of the trachea. Unlike standard (direct) laryngoscopes, they include a camera at the tip of the blade and display unit to provide an indirect view of the vocal cords (glottis). They are now routinely used for both standard and anticipated difficult tracheal intubation, and are recommended for difficult intubation in UK national guidelines.

Some videolaryngsocopes have a channel as a guide to help with placement of a tracheal tube and some are without a channel. The non-channelled videolaryngoscopes with acute-angled blades require a bougie or stylet to facilitate the passage of a tracheal tube through the glottis into the trachea.

One problem commonly encountered when using a standard bougie, is the tip of the bougie abutting on the anterior part of glottis and entrance to the windpipe (trachea) and not advancing further into the trachea. This is known as anterior impingement. This can increase the likelihood of repeated intubation attempts, failed intubation and airway trauma. C-Mac is a commonly used non-channelled videolaryngoscope and has been shown to have high first attempt success rate as compared to other videolaryngoscopes, however, the acute angled D-blade requires a bougie to facilitate tracheal intubation.

The recently introduced flexible tip bougie is likely to overcome the problem of anterior impingement, due to the ability to flex the tip in the posterior direction once the tip enters the glottis. Comparing the efficacy of these devices could help inform anaesthetists' decisions in the future when faced with a potentially difficult airway.

ELIGIBILITY:
Inclusion Criteria:

- Patients aged above 18, presenting for elective surgical procedures and requiring general anaesthesia tracheal intubation.

Exclusion Criteria:

* Patients who are do not want to take part or do not give consent
* Patients below 18 years of age
* Patient physical status of ASA 4 and 5,
* Patients deemed to require awake intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cyprian Mendonca, Phd, MD FRCA, Principal Investigator — University Hospitals Coventry & Warwickshire NHS Trust
Locations (1):
- University Hospitals Coventry & Warwickshire NHS Trust, Coventry, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Endotracheal Intubation With C-MAC D Blade Videolaryngoscopy and Standard Bougie | Endotracheal Intubation With C-MAC D Blade Videolaryngoscopy and Flexi-tip Bougie
Started | 80 | 80
Completed | 80 | 80 (completed)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Endotracheal Intubation With C-MAC D Blade Videolaryngoscopy and Standard Bougie | Endotracheal Intubation With C-MAC D Blade Videolaryngoscopy and Flexi-tip Bougie | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 69 | 70 | 139
  >=65 years | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: year] | 55.3 (16.3) | 55.2 (16.1) | 55.2 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 46 | 86
  Male | 40 | 34 | 74
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 80 | 80 | 160

OUTCOME MEASURES:

1. Primary Outcome: Modified Intubation Difficulty Scale Score (mIDS)
Description: Composite score of difficulty of tracheal intubation using the bougie devices minimum score is zero, maximum possible score is 10, higher values represent worse outcome. Total score is sum of sub scales, values are numbers Total 6 sub scale from N1 to N6 ( N1: 0-2, N2: 0-1, N3:0-5, N4: 0-1, N5 0-1, N6 0-1, so total mIDS score is sum of N1 to N 6 sub scales)
Time Frame: average 1 minute
Measure: Median (Inter-Quartile Range); unit: score on a scale range of 0 to 10 number
Arm/Group | Endotracheal Intubation With C-MAC D Blade Videolaryngoscopy and Standard Bougie | Endotracheal Intubation With C-MAC D Blade Videolaryngoscopy and Flexi-tip Bougie
Number analyzed (Participants) | 80 | 80
score on a scale range of 0 to 10 number | 1 [0 to 2] | 0 [0 to 1]

2. Secondary Outcome: Time to Successful Tracheal Intubation
Description: Time from when the videolaryngoscope is introduced into the oral cavity until the first capnography waveform is obtained.
Time Frame: less than two minutes
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Endotracheal Intubation With C-MAC D Blade Videolaryngoscopy and Standard Bougie | Endotracheal Intubation With C-MAC D Blade Videolaryngoscopy and Flexi-tip Bougie
Number analyzed (Participants) | 80 | 80
seconds | 42.9 (9.1) | 41.0 (6.1)

3. Secondary Outcome: Laryngoscopy Time
Description: Time from when the videolaryngoscope is introduced into the oral cavity to best view of the glottis (vocal cords).
Time Frame: less than one minute
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Endotracheal Intubation With C-MAC D Blade Videolaryngoscopy and Standard Bougie | Endotracheal Intubation With C-MAC D Blade Videolaryngoscopy and Flexi-tip Bougie
Number analyzed (Participants) | 80 | 80
seconds | 5 (2) | 4.6 (1.7)

4. Secondary Outcome: Overall First Attempt Success Rate
Description: This is the percentage of patients being successfully intubated at the first attempt. This will be compared for two bougies
Time Frame: average 1 minute
Measure: Count of Participants; unit: Participants
Arm/Group | Endotracheal Intubation With C-MAC D Blade Videolaryngoscopy and Standard Bougie | Endotracheal Intubation With C-MAC D Blade Videolaryngoscopy and Flexi-tip Bougie
Number analyzed (Participants) | 80 | 80
Participants | 79 | 80

5. Secondary Outcome: Anaesthetist's Visual Analogue Score for Ease of Use of the Bougie
Description: This is scored between 0 to 10, 0 being easy to use and 10 being extremely difficult to use
Time Frame: average 1 minute
Population: this data was not collected and therefore not analysed
Arm/Group | Endotracheal Intubation With C-MAC D Blade Videolaryngoscopy and Standard Bougie | Endotracheal Intubation With C-MAC D Blade Videolaryngoscopy and Flexi-tip Bougie
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 hours
Description: No adverse events
Arm/Group | Endotracheal Intubation With C-MAC D Blade Videolaryngoscopy and Standard Bougie | Endotracheal Intubation With C-MAC D Blade Videolaryngoscopy and Flexi-tip Bougie
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 0/80 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT04973176/Prot_000.pdf